CLINICAL TRIAL: NCT07076927
Title: Sagittal Radiographic Analysis of Spinopelvic and Coccygeal Alignment in Sitting and Standing Positions in Patients With Coccydynia
Brief Title: Sagittal Spinopelvic and Coccygeal Alignment in Sitting and Standing Positions in Coccydynia
Acronym: Coccydynia
Status: Completed | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aslinur Keles Ercisli, MD, PhD, Principal Investigator, Fatih Sultan Mehmet Training and Research Hospital
Other Study IDs: 2024/4-4/6
Record Dates: First submitted 2025-06-03; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Coccydynia; Sagittal Balance; Morphological Analysis and Classification
Keywords: Coccygeal morphometry; spinopelvic morphometry; os coccygis; sagittal plane; coccydynia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coccydynia: Coccydynia patients

SUMMARY:
This observational cross-sectional study aims to investigate the differences in spinopelvic and coccygeal morphometric parameters in standing and sitting positions among patients diagnosed with coccydynia. A total of 50 adult patients (aged 25-65 years) diagnosed with coccydynia based on clinical evaluation and imaging findings were included. Lateral radiographs were obtained in both standing and sitting positions. Radiological assessments included spinopelvic parameters such as sacral slope (SS), pelvic tilt (PT), pelvic incidence (PI), sacral table angle (STA), and sacral kyphosis (SK), along with coccygeal morphology based on the Postacchini-Massobrio classification. The study further aimed to explore whether these morphometric differences are associated with the presence of low back pain and to assess variations across different coccygeal morphology types.

DETAILED DESCRIPTION:
Coccydynia is a condition characterized by pain in the coccygeal region, often exacerbated by sitting and postural changes. While its etiology is multifactorial, anatomical variations in coccygeal and spinopelvic alignment may play a significant role in symptom development. Despite increasing attention to coccygeal mobility and morphology in radiological evaluations, the relationship between coccygeal type, spinopelvic alignment, and posture-specific morphometric changes has not been fully clarified.

This observational cross-sectional study was designed to evaluate morphometric parameters of the sacropelvic and coccygeal regions in both standing and sitting positions in patients diagnosed with coccydynia. The study included 50 adult patients (42 female, 8 male) aged between 25 and 65 years who were diagnosed with coccydynia based on clinical findings and radiological confirmation. Lateral radiographs were obtained in both weight-bearing and seated positions to allow for comparative measurement.

The following radiological parameters were assessed: thoracic kyphosis (TK), lumbar lordosis (LL), sagittal vertical axis (SVA), thoracopelvic angle and its modification (TPA-T1PA), sacral slope (SE), pelvic incidence (PI), pelvic tilt (PT), spinosacral angle (SSA), sacral table angle (STA), and sacral kyphosis (SK). Coccygeal features were evaluated based on vertebral segment number, sacrococcygeal and intercoccygeal joint fusion, segmental angulation, and mobility status. Morphological types were categorized using the modified Postacchini-Massobrio classification. The presence of coccygeal spicules and their frequency across types were recorded. Dynamic morphometric assessments included sacrococcygeal angle (SKA), intercoccygeal angle (IKA), coccygeal height (KY), sacral height (SY), and sacrococcygeal height (SKY). Mobility was determined by comparing the angular displacement between standing and sitting radiographs and classified as normal, hypermobile, hypomobile, or posterior luxation, depending on the flexion-extension response and translation under load.The study aimed to investigate the changes in these parameters between postures and explore whether these variations are associated with the presence of low back pain and functional impairment. Additionally, differences among coccygeal morphology subgroups in terms of spinopelvic parameters were analyzed.

ELIGIBILITY:
Inclusion Criteria:

Patients aged between 25 and 65 years

Clinically diagnosed with coccydynia

Provided informed consent to participate in the study

Exclusion Criteria:

Presence of any disease that may cause spinal malalignment

Any hip- or knee-related condition that may lead to spinal malalignment

History of surgery involving the cervical, thoracic, lumbar, or coccygeal spine

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients aged 25 to 65 years who presented to the University of Health Sciences Fatih Sultan Mehmet Training and Research Hospital with a preliminary diagnosis of coccydynia and were clinically confirmed were consecutively enrolled.
  Patients with a history of spinal trauma, surgery, congenital deformities, malignancy, or rheumatological disease were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-05-25 (Actual)

PRIMARY OUTCOMES:
Sacral Slope (SS) | At baseline (single time point)
  Sacral slope will be measured on standardized lateral radiographs in both standing and sitting positions.
Pelvic Tilt (PT) | At baseline (single time point)
  Pelvic tilt will be measured on sagittal radiographs in both standing and sitting positions.
Pelvic Incidence (PI) | At baseline (single time point)
  Pelvic Incidence will be measured on sagittal radiographs in both standing and sitting positions.
Spinosacral Angle (SSA) | At baseline (single time point)
  Spinosacral Angle will be measured on sagittal radiographs in both standing and sitting positions.
Sacral Kyphosis (SK) | At baseline (single time point)
  Sacral Kyphosis will be measured on sagittal radiographs in both standing and sitting positions.
Sacral Table Angle (STA) | At baseline (single time point)
  Sacral Table Angle will be measured on sagittal radiographs in both standing and sitting positions.
Thoracic Kyphosis (TK) | At baseline (single time point)
  Thoracic Kyphosis will be measured on sagittal radiographs in both standing and sitting positions.
Lumbar Lordosis (LL) | At baseline (single time point)
  Lumbar Lordosis will be measured on sagittal radiographs in both standing and sitting positions.
Sagittal Vertical Axis (SVA) | At baseline (single time point)
  Sagittal Vertical Axis will be measured on sagittal radiographs in both standing and sitting positions.
Thoracolumbar Angle (TPA-T1PA) | At baseline (single time point)
  Thoracolumbar Angle will be measured on sagittal radiographs in both standing and sitting positions.
Coccygeal Morphology- Vertebral Segment Number | At baseline (single time point)
  Coccygeal features will be evaluated
Coccygeal Morphology- sacrococcygeal joint fusion | At baseline (single time point)
  Coccygeal features will be evaluated
Coccygeal Morphology- intercoccygeal joint fusion | At baseline (single time point)
  Coccygeal features will be evaluated
Coccygeal Morphology- segmental angulation | At baseline (single time point)
  Coccygeal features will be evaluated
Coccygeal Morphology- presence of coccygeal spicules | At baseline (single time point)
  Coccygeal features will be evaluated
Coccygeal Morphometry Type | At baseline (single time point)
  Classification (Type 1-5)
Coccygeal Mobility | At baseline (single time point)
  Coccygeal mobility will be assessed by measuring the angular difference of the coccyx between the standing and sitting positions on lateral radiographs. The change in coccygeal angle reflects the degree of coccygeal movement during postural transition.
Sacrococcygeal Angle (SKA) | At baseline (single time point)
  SKA will be measured using the angle between the sacral axis and first coccygeal segment on lateral radiographs.
Intercoccygeal Angle (IKA) | At baseline (single time point)
  IKA will be measured as the angle between coccygeal segments
Coccygeal Height (KY) | At baseline (single time point)
  The vertical height of the coccyx from the tip to the base will be measured in the sagittal plane.
  ertical height of the coccyx from the tip to the base will be measured in the sagittal plane.
  Vertical height of the coccyx from the tip to the base will be measured in the sagittal plane.
Sacral Height (SY) | At baseline (single time point)
  Vertical sacral height will be assessed from the superior to the inferior sacral end on the lateral radiograph.
  ertical height of the coccyx from the tip to the base will be measured in the sagittal plane.
  Vertical height of the coccyx from the tip to the base will be measured in the sagittal plane.
Sacrococcygeal Height (SKY) | At baseline (single time point)
  Combined vertical height from sacral promontory to coccyx.

SECONDARY OUTCOMES:
Clinical Assessment- Pain severity | At baseline (single time point)
  Unit of Measure: Units on a Numeric Rating Scale (0-10) Description: Pain severity will be assessed using the Numeric Rating Scale (NRS), where 0 indicates no pain and 10 indicates the worst imaginable pain.
Clinical Assessment - Quality of Life (SF-12) | At baseline (single time point)
  Unit of Measure: SF-12 Score (0-100) Description: General health-related quality of life will be evaluated using the 12-Item Short Form Survey (SF-12).
Clinical Assessment - Disability - Oswestry Disability Index (ODI) Score | At baseline (single time point)
  Unit of Measure: Score (0-100)
  Description:
  Functional disability related to low back pain will be assessed using the Oswestry Disability Index (ODI). The ODI is a validated questionnaire consisting of 10 sections, each scored from 0 to 5. The total score is converted to a percentage, with higher scores indicating greater disability.

CONTACTS AND LOCATIONS:
Overall Officials: Aslinur Keles, MD., PhD, Principal Investigator — Fatih Sultan Mehmet Training and Research Hospital
Locations (1):
- Fatih Sultan Mehmet Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
undecided